CLINICAL TRIAL: NCT01919281
Title: High Intensity Interval Training or Strength Training in Women With Polycystic Ovary Syndrome. A Randomized Controlled Trial
Brief Title: High Intensity Interval Training or Strength Training in Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/886
Record Dates: First submitted 2013-07-17; First posted 2013-08-08 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: exercise; resistance training; insulin resistance; high intensity interval training
MeSH Terms: conditions — Polycystic Ovary Syndrome; Motor Activity; Insulin Resistance | interventions — Resistance Training; High-Intensity Interval Training; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- strength training (Experimental): The subjects will attend for supervised training three sessions per week for 10 weeks (9-12). The strength training program involves dynamic contraction at intensities of 60 - 70 % of 1 repetition maximum (RM) to improve strength and muscle hypertrophy. Each session will contain 8 exercises on the major muscle groups. Each drill consists of 10-12 repetitions (reps) x 3 sets separated by one minute rest between sets.
  Interventions: Behavioral: strength training
- interval training (Experimental): High intensity interval training (HIT) three times per week. The three weekly supervised HIT sessions will include two 4x4 min interval sessions and one 10x1 min session. The HIT consist of "uphill" treadmill running/walking.
  Interventions: Behavioral: interval training
- control (No Intervention): Based on the Norwegian recommendation we will encourage the control group to perform 60 minutes of physical activity at moderate to high intensity on a daily basis.

INTERVENTIONS:
Behavioral: strength training
  Other Names: resistance training
  Arms: strength training
Behavioral: interval training
  Other Names: high-intensity exercise; aerobic exercise
  Arms: interval training

SUMMARY:
The aim is to investigate whether strength training or high intensity interval training is effective in improving insulin sensitivity, cardiovascular outcomes, body composition and reproductive outcomes in women with Polycystic Ovary Syndrome (PCOS).

Few studies have examined the effect of strength training alone on insulin sensitivity, reproductive outcomes and body composition in women with PCOS. Most previous studies on aerobic exercise in PCOS have applied moderate exercise intensity.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age 18-45 years old
* PCOS

Exclusion Criteria:

* Regular high intensity endurance or strength training (two or more times per week of vigorous exercise).
* Concurrent treatments (insulin sensitizers or drugs known to affect gonadotropin or ovulation, with a wash out period of 1 months prior to inclusion).
* On-going pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
insulin resistance | 10 weeks
  measured with the homeostatic model assessment for insulin resistance (HOMA-IR) method

SECONDARY OUTCOMES:
Body composition | 10 weeks
  Measured as body fat % on an impedance scale and waist circumference
Maximum oxygen uptake | 10 weeks
  Measured during maximum effort exercise test
Endothelial function | 10 weeks
  Flow mediated dilatation of the brachial artery.

OTHER OUTCOMES:
Menstruation diary | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Trine Moholdt, phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of circulation and medical imaging , NTNU, Trondheim, Norway

REFERENCES:
- [Result] Almenning I, Rieber-Mohn A, Lundgren KM, Shetelig Lovvik T, Garnaes KK, Moholdt T. Effects of High Intensity Interval Training and Strength Training on Metabolic, Cardiovascular and Hormonal Outcomes in Women with Polycystic Ovary Syndrome: A Pilot Study. PLoS One. 2015 Sep 25;10(9):e0138793. doi: 10.1371/journal.pone.0138793. eCollection 2015. PMID 26406234